CLINICAL TRIAL: NCT03959462
Title: Supporting Decisions With Transcranial Direct Current Stimulation in Healthy Young and Elderly Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2017-01664; 17C195 (Other Grant/Funding Number: Novartis Foundation for medical-biological research)
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Real tDCS; Sham tDCS
Keywords: tDCS

STUDY DESIGN:
Intervention Model Description: Participants are allocated to one of 2 groups: real tDCS or sham.
Who Masked: Participant, Investigator
Masking Description: Double blind design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS (Experimental): 20 min of 1 mA real anodal transcranial direct current stimulation applied via 5x7 cm rubber electrodes over the DLPFC (current density: 0.028 mA/cm2). Additional ramp-up and ramp-down phase at beginning and end of stimulation lasting for 15 s. Electrodes remain attached to the participant's head for the duration of the decision task.
  Interventions: Device: real anodal transcranial direct current stimulation
- Sham tDCS (Sham Comparator): 30 s of 1 mA anodal tDCS applied via 5x7 cm rubber electrodes over the DLPFC (current density: 0.028 mA/cm2). Additional ramp-up and ramp-down phase at beginning and end of stimulation lasting for 15 s. Electrodes remain attached to the participant's head for the duration of the decision task.
  Interventions: Device: sham transcranial direct current stimulation

INTERVENTIONS:
Device: real anodal transcranial direct current stimulation — A neuroConn DC-Stimulator PLUS (neuroCare Group, Ilmenau, Germany) will be used.
  Arms: Real tDCS
Device: sham transcranial direct current stimulation — A neuroConn DC-Stimulator PLUS (neuroCare Group, Ilmenau, Germany) will be used.
  Arms: Sham tDCS

SUMMARY:
Decisions are part of the daily life. On the neuronal level, activity in the dorsolateral prefrontal cortex (dlPFC) is important during complex decisions (e.g., whether something is emotional for a person or not). We apply transcranial direct current stimulation (tDCS) with the aim to increase dlPFC activity and thereby modulate decisions towards emotional content.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Non-smokers
* Right-handedness
* Native German speakers or comparable level of fluency
* Normal or corrected-to-normal vision

Exclusion Criteria:

* Neurological or psychiatric condition (other than diagnosed cognitive impairment)
* Past head injuries
* Magnetizable implants
* History of seizures
* Current or life-time alcohol or drug abuse
* Skin diseases
* tES in the 3 months preceding or during the present study
* Caffeine 3 hours prior to training

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 254 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Influence of Stimulation on the Decisions | 10 minutes
  Number of words which were rated as positive or negative.

SECONDARY OUTCOMES:
Profile of Mood States (POMS; before stimulation) | 3 minutes
  Changes in the subjective measure mood, assessed with questionnaire Scores for each item is recorded as 0 for "not at all" up to 6 for "very strong". A Total Mood Disturbance (TMD) score is calculated by summing the totals for the negative subscales dejection (14 items), fatigue (7 items) and discontent (7 items) and then subtracting the total for the positive subscale zest (7 items).
Profile of Mood States (POMS; after stimulation) | 3 minutes
  Changes in the subjective measure mood, assessed with questionnaire Scores for each item is recorded as 0 for "not at all" up to 6 for "very strong". A Total Mood Disturbance (TMD) score is calculated by summing the totals for the negative subscales dejection (14 items), fatigue (7 items) and discontent (7 items) and then subtracting the total for the positive subscale zest (7 items).
Positive and Negative Affect Schedule (PANAS; before stimulation) | 2 minutes
  Changes in the subjective measure mood, assessed with self-report questionnaire divided into two mood scales. One scale measures a person's positive emotion and the other scale measures the negative. Each segment has ten terms, which can be rated on a scale of 1 to 5 to indicate the extent to which the respondent agrees that this applies to him (higher values means higher agreement).
Positive and Negative Affect Schedule (PANAS; after stimulation) | 2 minutes
  Changes in the subjective measure mood, assessed with self-report questionnaire divided into two mood scales. One scale measures a person's positive emotion and the other scale measures the negative. Each segment has ten terms, which can be rated on a scale of 1 to 5 to indicate the extent to which the respondent agrees that this applies to him (higher values means higher agreement).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Peter, PD, Principal Investigator — Universitäre psychiatrische Dienste Bern (UPD), University of Bern
Locations (1):
- Klinik für Alterspsychiatrie und Psychotherapie UPD Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No